CLINICAL TRIAL: NCT00298090
Title: An Evaluation of a Radial Arterial Line's Effect on StO2 Monitoring Using the InSpectra® Tissue Spectrometer
Brief Title: Evaluation of a Radial Arterial Line's Effect on StO2 Monitoring
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Other Study IDs: 045-1502-319; 045-1502-319 (Other: Institutional Review Board)
Record Dates: First submitted 2006-02-27; First posted 2006-03-01 (Estimated); Results first posted 2013-08-02 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Oxygenation
Keywords: Oxygenation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- StO2 values: StO2 monitoring
  Interventions: Device: StO2 monitoring

INTERVENTIONS:
Device: StO2 monitoring — placement of the StO2 device/ external noninvasive
  Other Names: external near infrared spectroscopy

SUMMARY:
Measuring tissue oxygen saturation (St02) in the thenar eminence is emerging as a measurement of resuscitation. However, no study to our knowledge has evaluated the effects of an arterial line in the radial artery supplying this muscle bed on St02. This study will attempt to address the interaction between an arterial line and St02 monitoring in the thenar eminence. As most patients who require aggressive resuscitation will have an arterial line, it is important to understand what if any impact this will have on St02 in the same extremity.

ELIGIBILITY:
Inclusion Criteria:

* Standard of care placement of arterial line
* 18 years of age or older

Exclusion Criteria:

* Pregnant females
* Nursing mothers
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients wiht arterial lines
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2006-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lopez P Peter, M.D., Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- University Hospital, San Antonio, Texas, United States

REFERENCES:
- See also: device information — http://www.htibiomeasurement.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from inpatients at a local hospital's Intensive Care Unit (ICU)
Groups:
- StO2 Values Pre and Post Arterial Line Placement: single arm study of StO2 in subjects undergoing placement of arterial line. Measurements of StO2 will be taken before and after arterial line placement.
Period: Overall Study
Arm/Group | StO2 Values Pre and Post Arterial Line Placement
Started | 47
Completed | 29 (Eighteen subjects were not included in final analysis due to incomplete data sets)
Not Completed | 18

BASELINE CHARACTERISTICS:
Groups:
- StO2 Values: StO2 values pre and post arterial line placement.
Arm/Group | StO2 Values
Number analyzed (Participants) | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 47
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 28
Region of Enrollment [Number; unit: participants]
  United States | 47

OUTCOME MEASURES:

1. Primary Outcome: Tissue Oxygen Saturation (StO2) Measurement on the Extremity With a Radial Arterial Line
Description: Using near-infrared spectroscopy, the external device recorded raw StO2 values every 3.5 seconds for approximately 5 minutes prior to and immediately following the insertion of a radial arterial catheter on the ipsilateral side. The raw values were then compiled into one-minute averages.
Time Frame: up to 15 minutes
Population: Data from 18 subjects not used due to only partial data captured resulting from logistical issues.
Measure: Mean (95% Confidence Interval); unit: StO2 percent saturation
Groups:
- StO2 Values: StO2 pre and post catheter placement
Arm/Group | StO2 Values
Number analyzed (Participants) | 29
StO2 percent saturation | 0.68 [-0.80 to 1.48]
Statistical Analysis 1: Comparison: StO2 Values; Test type: Superiority or Other; p = 0.55, repeated measures model; Other = 0, 95% CI 2-sided [-0.80 to 1.48] — A repeated measures model was used to assess whether the one-minute average StO2 values differed systematically between pre and post arterial line placement

ADVERSE EVENTS:
Time Frame: During StO2 measurement, up to 15 minutes
Description: No adverse events observed. 47 subjects enrolled, 29 subjects completed. Non invasive StO2 measurement device used to obtain values. No adverse events occured during the course of subjects participation.
Groups:
- StO2: StO2 measurements pre and post arterial line catheter placement.
Arm/Group | StO2
Serious Adverse Events (participants affected / at risk) | 0/47
Other Adverse Events (participants affected / at risk) | 0/47

LIMITATIONS AND CAVEATS:
Eighteen subjects were not included in final analysis due to incomplete data sets; unsuccessful arterial line placement, technical problems in applying StO2 device, unreliable data or partial data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes